CLINICAL TRIAL: NCT02377440
Title: Effects of Angiotensin Converting Enzyme Inhibitors (ACEI) on Bone Turnover
Brief Title: Effects of ACEI on Bone Turnover
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nahid Rianon, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-13-0634
Record Dates: First submitted 2014-03-19; First posted 2015-03-03 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Bone Turnover Status in Hypertensive Patients
Keywords: ACE inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that older persons (≥45 years) treated with ACEI for HTN control will have: i) improved status of bone turnover (decreased P1NP and CTX), and ii) decreased levels of RANKL and RANKL/OPG, compared to those not treated with ACEI and not using RAS-related medications

ELIGIBILITY:
Inclusion Criteria:

* at least 45 years of age
* a diagnosis of (either new or uncontrolled) HTN who will need a new medication for HTN control
* able to consent (no medial issues impairing judgment for consenting based on clinical providers' judgment).

Exclusion Criteria:

* younger than 45 years of age
* a diagnosis of metabolic bone disease
* a diagnosis of osteoporosis or use of medication to treat osteoporosis
* a diagnosis of diabetes mellitus, or renal insufficiency, or cancer
* history of allergy to ACEI or ARB, 6) history of use of ACEI or ARB.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 60 patients (30 men and 30 women) 45 years or older will be recruited at designated outpatient clinics and randomly allocated 1:1 to receive ACEI vs. a non RAS-related antihypertensive medication.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in serum CTX levels in pg/mL | baseline, 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nahid Rianon, MD, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas